CLINICAL TRIAL: NCT06637046
Title: Is the Phoenix Sign Phenomenon Due to Vasodilation? a Double-Blinded, Randomized Controlled Trial Comparing Motor Function Recovery After Diagnostic Common Fibular Nerve Block with Lidocaine and Papaverine
Brief Title: Does Blood Vessel Vasodilation, Caused by Focal Infiltration of Lidocaine Cause Temporary Nerve Functional Recovery for Patients with Common Peroneal Nerve Injury or Entrapment: Testing the 'Phoenix Sign' Effect Between Lidocaine (a Common Local Anesthetic) and Papaverine, a Know Vasodilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Barrett (Other)
Collaborators: US Neuropathy Centers (Other)
Responsible Party: Sponsor-Investigator, Stephen Barrett, CEO US Neuropathy Centers Medical Director, US Neuropathy Centers
Organization: US Neuropathy Centers (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Study 20-391
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Drop Foot
Keywords: Drop Foot; Common Peroneal Nerve Palsy; Weakness of Anterior and Lateral Compartment of Leg
MeSH Terms: conditions — Peroneal Neuropathies | interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lidocaine group (Experimental): Patients randomized to this arm received less than a .5cc infiltration of plain lidocaine
  Interventions: Diagnostic Test: Diagnostic procedures; Diagnostic Test: Lidocaine HCl
- Papavarine (Experimental): Patients randomized to this arm received less than a .5cc infiltration of 10mg/ml papaverine
  Interventions: Diagnostic Test: Diagnostic procedures; Diagnostic Test: Lidocaine HCl

INTERVENTIONS:
Diagnostic Test: Diagnostic procedures — A 30-gauge 1-inch needle was inserted adjacent to, but not within, the CFN. The infiltrate was delivered at the level of the fibular neck just proximal to where the CPN coursed beneath the deep fascia of the peroneus longus. This was immediately adjacent to the first known anatomical site of compression of the CPN. 0.3cc of the drug was delivered.
Diagnostic Test: Lidocaine HCl — This study compares the vasodilatory effects of lidocaine to papaverine after diagnostic infiltration of the Common Peroneal Nerve in patients with demonstrated motor weakness of the EHL (extensor hallucis longus).
  Other Names: Papaverine

SUMMARY:
The goal of this clinical trial is to compare lidocaine without epinephrine to papaverine a known vasodilatory agent, in creating improved motor strength in patients with drop foot involving an entrapment of the Common Peroneal Nerve. This phenomenon has been named the Phoenix Sign and is a very specific peripheral nerve block.

Researchers will compare the effects of the above agent for pre and post infiltration changes in motor strength.

Participants will:

* Will be randomized to one of either agents already listed
* After receiving the ultrasound guided injection, motor testing will be evaluated in 4-6 minutes with manual motor strength testing of the anterior compartment muscles.
* No additional follow will be required

DETAILED DESCRIPTION:
A double-blinded, randomised, prospective controlled trial was conducted at US Neuropathy Centers in Marietta, GA, under the approval of the Kennesaw State University Institutional Review Board. Patients with weak dorsiflexion of the ankle or a drop foot were recruited from the existing clinical practice at US Neuropathy Centers. Cohort inclusion criteria also included a stable medical and medication status, ages 18-85, speaking English as the primary language, and ambulatory. Walking aids or ankle-foot orthosis were permitted.. Based on the inclusion criteria, only 20 patients were enrolled. Patients were recruited over a period of 1 year and two months from January 2021 to March 2022 with no requirement for follow-up. The enrolment phase was concluded as the study was originally designed as a pilot investigation, with recruitment limited to a single, small medical practice. A total of 20 patients were successfully enrolled within this setting.Participants were randomised by the throw of dice to injection of 0.3 cc of Papaverine HCl 10 mg/mL or 0.3 cc of 1% Lidocaine HCl adjacent to CFN in a room separate from patient room. Injection solutions were prepared by non-blinded assistants and were visually indistinguishable. Patients and physicians are blinded to drugs received. Motor strength of the Extensor Hallucis Longus (EHL), Tibialis Anterior (TA), and Extensor Digitorum Longus (EDL) muscles were tested. Strength was rated according to the Medical Research Council Manual Muscle Testing scale 0-5. The CFN at the fibular neck was identified under high-resolution ultrasound imaging. The injection site was prepared with alcohol, and ethyl chloride was used to anaesthetise the skin. A 30-gauge 1-inch needle was inserted adjacent to, but not within, the CFN. The infiltrate was delivered at the level of the fibular neck just proximal to where the CPN coursed beneath the deep fascia of the peroneus longus. This was immediately adjacent to the first known anatomical site of compression of the CPN. 0.3cc of the drug was delivered.

The investigator then waited approximately five minutes and re-tested motor strength of the Extensor Hallucis Longus (EHL), Tibialis Anterior (TA), and Extensor Digitorum Longus (EDL) muscles manually.

ELIGIBILITY:
Inclusion Criteria:Cohort inclusion criteria also included a stable medical and medication status, ages 18-85, speaking English as the primary language, and ambulatory. Walking aids or ankle-foot orthosis were permitted.

-

Exclusion Criteria: Patients with normal motor strength of the anterior compartment of the leg.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Manual Motor Strength Testing of Anterior Compartment | From enrollment to evaluation which is complete upon the first study visit after infiltration of the agents. The increased motor effect after infiltration is only apparent for 10 minutes or less
  Motor strength of the Extensor Hallucis Longus (EHL), Tibialis Anterior (TA), and Extensor Digitorum Longus (EDL) muscles were tested. Strength was rated according to the Medical Research Council Manual Muscle Testing scale 0-5.

CONTACTS AND LOCATIONS:
Locations (1):
- US Neuropathy Centers, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowley MP, Doughty CT. Entrapment Neuropathies of the Lower Extremity. Med Clin North Am. 2019 Mar;103(2):371-382. doi: 10.1016/j.mcna.2018.10.013. Epub 2018 Dec 3. PMID 30704688
- [Derived] Barrett SL, Boyd B, DuCasse S, Nassier W, Mitchell N, Nagra AP, Dalmau-Pastor M, Yamasaki DS, Nickerson S. Is the phoenix sign phenomenon due to vasodilation? A double-blinded, randomized controlled trial comparing motor function recovery after diagnostic common fibular nerve block with lidocaine and papaverine. BMC Musculoskelet Disord. 2024 Oct 23;25(1):840. doi: 10.1186/s12891-024-07972-3. PMID 39443927